CLINICAL TRIAL: NCT05746689
Title: Combination Therapy of Sirolimus and Glucocorticoids for the Maintenance of Remission in Patients With IgG4-related Disease
Brief Title: Study of Sirolimus in IgG4-related Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University International Hospital (Other)
Responsible Party: Principal Investigator, Yu Ying Wang, Principal Investigato, Peking University International Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sirolimus for IgG4-RD
Record Dates: First submitted 2023-02-13; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: IgG4-related Disease
Keywords: IgG4-related disease; sirolimus; mTOR
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Sirolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- glucocorticoid and sirolimus combination therapy (Experimental): Prednisone acetate 0.8mg/Kg/d (maximum dose 60mg/d), reduced by 5mg every 14 days, reduced by 2.5mg every 2 weeks after 30mg/d until discontinuation. At the same time, treatment for prevention or control of osteoporosis was given.
  Sirolimus: 2mg/day for the first three days and 1mg/day thereafter. The plasma drug concentration was monitored at 14 days, 12 weeks, and 48 weeks of medication to maintain a plasma drug concentration of 4-15 ug/L.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus The efficacy is evaluated at 12 weeks, and treatment will be adjusted according to the control of disease and adverse effects.For experimental group, if a patient is assessed as treatment failure (TS), the patient should be withdrawn from the study and receive rescue treatment. Whereas, a patient would be transferred to the control group if he/ she cann't stand the side effects of sirolimus but not serious adverse event (SAE).
  Other Names: Prednisone

SUMMARY:
gG4-related disease (IgG4-RD) is a newly recognized systemic autoimmune disease that can involve the pan-creatobiliary tract, retroperitoneum/aorta, head and neck region, and salivary glands, et al. Glucocorticoids are the first-line agents for the treatment of IgG4-RD, however, in order to maintain long-term disease stability and avoid disease relapse, glucocorticoids maintenance therapy should last for a long period, which may induce various glucocorticoid-associated adverse reactions. Sirolimus plays dual roles in inhibiting lymphocyte activation and fibroblast proliferation. It is inferred from its mechanism that sirolimus is a good potential treatment option for IgG4-RD. Therefore, we conducted this single-arm clinical trial on patients with IgG4-RD to determine the efficacy and safety of sirolimus.

DETAILED DESCRIPTION:
IgG4-related disease (IgG4-RD) is a newly recognized systemic autoimmune disease that can involve the pan- creatobiliary tract, retroperitoneum/aorta, head and neck region, and salivary glands, et al. IgG4-RD is characterized by elevated serum IgG4 levels, tumefactive lesions with a dense lymphoplasmacytic infiltration rich in IgG4 positive plasma cells and storiform fibrosis of related organs.

Glucocorticoids are the first-line agents for the treatment of IgG4-RD, however, in order to maintain long-term disease stability and avoid disease relapse, glucocorticoids maintenance therapy should last for a long period, which may induce various glucocorticoid-associated adverse reactions. For some mild IgG4-RD patients without internal organ damage, long-term glucocorticoids therapy may have a low benefit/risk ratio. Further, a substantial proportion of patients cannot tolerate glucocorticoids.

Sirolimus, also known as rapamycin, is a macrolide compound that inhibits its mechanistic target (mTOR), which regulates cell growth and metabolism in response to environmental cues. mTOR is also essential in driving abnormal lineage specification within the immune system in various rheumatic diseases. We discovered that mTOR was highly activated in IgG4RD tissues, and its inhibitor sirolimus appeared as a good treatment candidate.

ELIGIBILITY:
Inclusion criteria:

1. Patients diagnosed with IgG4-RD according to the 2011 Comprehensive Diagnostic Criteria for IgG4-RD;
2. Status classified as active disease based on an IgG4-RD Responder Index (RI) ≥2 at screening.

1.Exclusion criteria: 2.Having used glucocorticoids (equivalent to more than 10mg per day of prednisone), immunosuppressant or biologic within 3 months prior to enrollment; 3.Having any contraindication of glucocorticoids or sirolimus, or allergy to sirolimus, or having experienced serious adverse reactions from previous use of any of the above drugs; 4.Combined with other connective disease; 5.History or evidence of a clinically unstable/uncontrolled disorder, condition or disease (including but not limited to cardiopulmonary, oncologic, renal, hepatic, metabolic, hematologic or psychiatric) other than IgG4-RD that, in the opinion of the Investigator, would pose a risk to patient safety or interfere with the study evaluation, procedures or completion; 6.Active infection, including hepatitis B virus, hepatitis C virus, and tuberculosis; 7.Malignancy within 5 years; 8.Other serious complications or general conditions do not permit; 9.Pregnancy or to be pregnant, or breast feeding; 10.Unable to adhere to follow-up or the patient refuses to provide consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PrRelapse rate | through study completion, an average of 1 year
  For patients who achieve disease response at 12 weeks, recurrence is defined as increases in the IgG4-RD RI ≥2 and/or the need for the reinstitution of treatment.

SECONDARY OUTCOMES:
Disease response rate at 12 weeks | 12 weeks of treatment
  Disease response is defifined as an improvement of the IgG4-RD RI ≥2 compared with baseline.
Remission rate at 48 weeks | 48 weeks of treatment
  Remission is defined as the achievement of an IgG4-RD RI of 0
Improvement of patient's global assessment (PGA) | 48 weeks of treatment
  PGA is a validated visual analogue scale that is scored by placing a vertical mark along a 100 mm horizontal line. Zero millimetre indicates no disease activity. A mark of 100 mm indicates the most active disease possible

CONTACTS AND LOCATIONS:
Overall Officials: Yuying Wang, Principal Investigator — Peking University International Hospital

IPD SHARING:
Plan to Share IPD: No